CLINICAL TRIAL: NCT00433641
Title: Pharmacogenomics of Weight Loss With Sibutramine in Obese and Overweight Patients
Brief Title: Weight Loss in Response to Sibutramine (MERIDIA) is Influenced by the Inherited Genes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Michael Camilleri, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-003371; NIH DK67071
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Obesity
Keywords: obesity; pharmacogenetics; sibutramine; adrenergic; serotonergic; body composition; gastric emptying
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): placebo tablet
  Interventions: Drug: sibutramine
- 2 (Experimental): sibutramine
  Interventions: Drug: sibutramine
- 3 (Experimental): sibutramine
  Interventions: Drug: sibutramine

INTERVENTIONS:
Drug: sibutramine — placebo
  Other Names: meridia
  Arms: 1
Drug: sibutramine — oral 15 mg sibutramine once per day
  Other Names: MERIDIA
  Arms: 3
Drug: sibutramine — oral sibutramine 10 mg once per day
  Other Names: MERIDIA
  Arms: 2

SUMMARY:
Control of food intake, size and frequency of meals are critical to the development of obesity. The stomach signals feelings of fullness after a meal and therefore plays a role in control of calorie intake. It is unclear whether the approved appetite reducing drug sibutramine changes the function of the stomach. Differences in the way individuals respond to treatment with the appetite suppressant sibutramine may also explain why some people lose weight while others do not.

In a previous study of 48 overweight or obese participants, we preliminarily observed that variation in the gene for the promoter of the serotonin transporter protein was significantly associated with degree of weight loss.

This new single center clinical study aims to evaluate the effects of the FDA-approved appetite suppressing medication, sibutramine (MERIDIA)on weight loss and stomach emptying in patients who are overweight or obese. The effect of individual differences in inherited genes that modify serrotonin and noradrenergic receptors on weight reduction with sibutramine will be tested.

DETAILED DESCRIPTION:
Background:. Genetic variations are potentially key to inter-individual differences in responses to treatment with the appetite suppressant sibutramine.

Overall Aims: To evaluate influence of genetic variation in candidate adrenergic and serotonergic control mechanisms on weight loss and gastric emptying response to sibutramine in obesity.

Methods: 180 overweight or obese (respectively BMI of 25-29.9 or 30 kg/m2) people treated with sibutramine (10 or 15 mg/day) or placebo for 12 wks. We shall collect DNA from venous blood sample at study entry, and use SERT-P genotype at baseline to stratify patients according to LL vs LS/SS genotype in both obese and overweight groups. The primary outcome measurement will be the association of clinical response (weight loss) and the influence of SERT-P and 2-MSP variation. A secondary outcome for descriptive purposes is the gastric emptying response to sibutramine treatment. Gastric emptying of solids will be measured using stable isotope method.

Anticipated Results: SERT-P genotype is significantly associated with the magnitude of weight loss in obese and overweight individuals.

Significance: Our study will provide the first evidence of the pharmacogenomic effects of sibutramine on weight loss in obesity and appraise the association of weight loss with change in gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight, overweight and obese subjects with BMI> 18 Kg/m2 residing in Olmsted County, MN: Otherwise healthy individuals who are not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrine (other than hyperglycemia not requiring medical therapy) and unstable psychiatric disease.
* Age: 18-65 years
* Gender: Men or women. Women of childbearing potential will have negative pregnancy test within 48 h of enrollment and before each radiation exposure.

Exclusion Criteria:

* Weight exceeding 300 pounds or 137 kilograms (due to limitations regarding SPECT imaging studies).
* Abdominal surgery other than appendectomy, Caesarian section or tubal ligation.
* Positive history of chronic gastrointestinal diseases, systemic disease that could affect gastrointestinal motility or use of medications that may alter gastrointestinal motility, appetite or absorption e.g., orlistat (Xenical).
* Significant psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Scale [HADS] self-administered alcoholism screening test (substance abuse) and the questionnaire on eating and weight patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a HADS score >8 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* Intake of medication, whether prescribed or OTC medication (except multivitamins) within 7 days of the study. Exceptions are birth control pill, estrogen replacement therapy, and thyroxine replacement.
* Concomitant use of MAOI inhibitors and other centrally acting appetite suppressants (since this would make them ineligible for sibutramine treatment).
* Hypersensitivity to sibutramine (since this would make them ineligible for sibutramine treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Association of weight loss with candidate genotypes | 2006-2007

SECONDARY OUTCOMES:
T1/2 gastric emptying of solids | 2006-2007
body composition (fat) | 2006-2007

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Camilleri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Grudell AB, Sweetser S, Camilleri M, Eckert DJ, Vazquez-Roque MI, Carlson PJ, Burton DD, Braddock AE, Clark MM, Graszer KM, Kalsy SA, Zinsmeister AR. A controlled pharmacogenetic trial of sibutramine on weight loss and body composition in obese or overweight adults. Gastroenterology. 2008 Oct;135(4):1142-54. doi: 10.1053/j.gastro.2008.07.009. Epub 2008 Jul 16. PMID 18725220